CLINICAL TRIAL: NCT04926493
Title: Structural and Microbiological Characterization of Endotracheal Tube Biofilm in Patients at Increased Risk for the Development of Ventilator-associated Pneumonia in the Intensive Care Unit
Acronym: BIOPAVIR
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: QUENOT-Maldiney 2021
Record Dates: First submitted 2021-05-27; First posted 2021-06-15 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Biofilm Formation; Structural and Microbiological Characterization of Endotracheal Tube Biofilm; Ventilator-associated Pneumonia (VAP)
MeSH Terms: conditions — Pneumonia, Ventilator-Associated

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- BIOPAVIR Cohort: Critically ill patient > 18 years of age with mechanical ventilation for >2 calendar days, at increased risk for the development of Ventilator-Associated Pneumonia in the Intensive Care Unit during COVID-19 pandemic.
  Interventions: Biological: microbiological characterization

INTERVENTIONS:
Biological: microbiological characterization — microbiological characterization of endotracheal tube biofilm

SUMMARY:
Ventilator-associated pneumonia (VAP) remains the most frequent healthcare-associated infection (HAI) in the intensive care unit (ICU) and one of the most critical risk factors associated with both significant morbidity as well as mortality. Although VAP treatment relies on early and appropriate antimicrobial therapy, several preventive measures have been described in the literature in order to limit its incidence and clinical impact in the ICU. Among these, preventing biofilm formation on the inner surface of the endotracheal tube appears to hold promise. Yet there is a lack of clinical relevant data documenting a causal relation between biofilm formation and VAP. Designed to overcome this critical limitation, the BIOPAVIR study intends to provide a better structural and microbiological characterization of endotracheal tube biofilm in critically ill patients at increased risk for the development of VAP in ICU during COVID-19 pandemic.

ELIGIBILITY:
Inclusion Criteria:

* patient > 18 years of age with mechanical ventilation for >2 calendar days

Exclusion Criteria:

* inability to collect or dispatch the endotracheal tube for proper characterization within 24 hours post-extubation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patient > 18 years of age with mechanical ventilation for >2 calendar days
Sampling Method: Non-Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
Development of Ventilator-associated pneumonia (VAP) | Immediately after extubation of the patient
  Provide a better understanding of the correlation between structural and microbiological characterization of endotracheal tube biofilm in critically ill patients and increased risk for the development of VAP in ICU during COVID-19 pandemic.

SECONDARY OUTCOMES:
Development of other VAP, healthcare-associated infection (HAI) or mortality | Immediately after extubation of the patient
  Provide a better understanding of the correlation between structural and microbiological characterization of endotracheal tube biofilm in critically ill patients and increased risk for the development of other VAP, healthcare-associated infection (HAI) or mortality in ICU during COVID-19 pandemic.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Dijon Bourgogne, Dijon, France

REFERENCES:
- [Result] Maldiney T, Pineau V, Neuwirth C, Ouzen L, Eberl I, Jeudy G, Dalac S, Piroth L, Blot M, Sautour M, Dalle F, Abdulmalak C, Ter Schiphorst R, Pugliesi PS, Poussant T, Ogier-Desserrey A, Fournel I, de Giraud d'Agay M, Jacquier M, Labruyere M, Aptel F, Roudaut JB, Vieille T, Andreu P, Prin S, Charles PE, Hamet M, Quenot JP. Endotracheal tube biofilm in critically ill patients during the COVID-19 pandemic : description of an underestimated microbiological compartment. Sci Rep. 2022 Dec 27;12(1):22389. doi: 10.1038/s41598-022-26560-w. PMID 36575298